CLINICAL TRIAL: NCT03346577
Title: Endovascular Treatment of Peripheral Artery Disease
Acronym: PAD
Status: Terminated | Type: Observational
Why Stopped: Termination of collaboration
Sponsor: be Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BM-PAD-01
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Peripheral Arterial Disease; Iliac Artery Disease; Below-the-knee Obstruction; Femoropopliteal Occlusive Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Stents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with peripheral artery disease: located in the common and external iliac artery, the common and superficial femoral artery, the popliteal artery and/or the below-the-knee (BTK) arteries (anterior tibial artery, posterior tibial artery or peroneal artery).
  Interventions: Device: stent or balloon

INTERVENTIONS:
Device: stent or balloon — Endovascular treatment with stent or balloon according to current practice
  Other Names: Optimed Sinus Superflex 635 stent; Cardionovum Legflow balloon; Optimed Nylotrack .035 + .018 balloons

SUMMARY:
The purpose of this observational study is to evaluate the performance and safety of endovascular treatment with stenting (Optimed Sinus Superflex 635) or balloon angioplasty (Cardionovum Legflow or Optimed Nylotrack .035 + .018) according to current practice. The goal of the study will be achieved by assessing binary restenosis with duplex ultrasound, peri- and postoperative complications, technical success, target lesion revascularization, amputation and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must sign the informed consent form prior to the index-procedure.
2. Patient is older than 18 years.
3. Patient is compliant with the requested follow-up visits at week 6 and month 12 and the treatment regime.
4. Patient suffers from intermittent claudication (Rutherford 2-3) or critical limb ischemia (Rutherford 4-5).
5. Target lesion is an occlusion or diameter stenosis is ≥70% by visual estimate.
6. Target lesion is located in the common and external iliac artery, in the common and superficial femoral artery, popliteal artery and/or the below-the-knee (BTK) arteries (anterior tibial artery, posterior tibial artery or peroneal artery) .

Exclusion Criteria:

1. Patients with Rutherford 0, 1 and 6.
2. Patient is pregnant.
3. Patients with serum creatinine >2.0 mg/dL or renal dialysis.
4. Patient has an acute thrombus or aneurysm in the target arteries.
5. Patient has a life expectancy of <12 months.
6. Patient with bypass that involves the target arteries.
7. Patient has a target lesion that cannot be crossed with a guidewire.
8. Patient suffers from acute limb ischemia defined as any sudden decrease in limb perfusion causing a potential threat to limb viability.
9. Patient has scheduled elective non-vascular procedures within 3 months after index-procedure. Vascular procedures are allowed within 3 months after the index-procedure if it is guaranteed that acetylic salicylic acid and clopidogrel intake is not interrupted.
10. Contraindication for anti-thrombotic therapy (coagulopathy, …).
11. Patient has a known intolerance to anti-thrombotic medication or contrast agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with peripheral artery disease, located in the common and external iliac artery, the common and superficial femoral artery, the popliteal artery and/or the below-the-knee (BTK) arteries (anterior tibial artery, posterior tibial artery or peroneal artery).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-05-02 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Binary restenosis | at 12 months follow-up
  Binary restenosis defined as ≥ 50% re-obstruction of the target lesion will be assessed by duplex ultrasound (peak systolic ratio >2.4)

SECONDARY OUTCOMES:
Device-related complications | up to 12 months follow-up
  Registration of peri- and early/late postoperative complications
Immediate procedural outcome | up to 12 months follow-up
  The combination of technical success defined as a successful access and deployment of the device and achievement of a final residual diameter stenosis of <30% of the treated target lesion on the procedural completion angiography.
  and procedural success defined as a combination of technical success and absence of procedural complications.
Clinical outcome | at baseline
  Rutherford classification
Clinical outcome | at 6 weeks follow-up
  Rutherford classification
Clinical outcome | at 12 months follow-up
  Rutherford classification
Primary sustained clinical improvement | at 12 months follow-up
  defined as sustained upward shift of ≥ 1 category on Rutherford classification without the need for repeated TLR in surviving patients.
Secondary sustained clinical improvement | at 12 months follow-up
  defined as sustained upward shift of ≥ 1 category on Rutherford classification including the need for repeated TLR in surviving patients.
Target lesion revascularization (TLR) | up to 12 months follow-up
  defined as an endovascular or surgical treatment due to a problem arising from the lesion (+1cm proximally and distally to include edge phenomena).
Mortality | up to 12 months follow-up
  Procedure-related and all-cause mortality.
Amputation | up to 12 months follow-up
  minor amputation defined as below the ankle and major defined as above the ankle.
Stent fracture | up to 12 months follow-up
  Only if restenosis occurs, stent fracture will be examined (when Optimed Sinus Superflex 635 stent is used).

CONTACTS AND LOCATIONS:
Locations (1):
- Mariaziekenhuis Noord-Limburg, Overpelt, Limburg, Belgium